CLINICAL TRIAL: NCT05016466
Title: GOLD 0 - DLCO 1: A Look Beyond the Obstruction. Is Spirometry Enough for COPD Screening?
Brief Title: GOLD 0 - DLCO 1: A Look Beyond the Obstruction. Is Spirometry Enough for COPD (Chronic Obstructive Pulmonary Disease) Screening?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: GOLD 0-DLCO 1
Record Dates: First submitted 2021-07-26; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: COPD, Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I. Patients with DLCO <80%.: Patients with DLCO <80% will be followed at baseline and once a year during the study
  Interventions: Other: Standard Care plus oxidative stress study plus inflammation biomarkers study
- Group II. Patients with DLCO ≥ 80%.: Patients with DLCO ≥80% only will be followed at baseline and year 5.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Standard Care — Patients will followed during 5 years, and only 2 visits , baseline and 5 years
  Groups: Group II. Patients with DLCO ≥ 80%.
Other: Standard Care plus oxidative stress study plus inflammation biomarkers study — Patients will followed during 5 years, Annual follo-up visits will be carried out during this period
  Groups: Group I. Patients with DLCO <80%.

SUMMARY:
This is a multicenter observational prospective study in smokers or ex-smokers with cumulative exposure ≥ 10 a / p (years / pack) with respiratory symptoms and presenting a normal spirometry.

The patients who sign the corresponding informed consent, will undergo a DLCO and will be divided into two groups according to the result:

* Group I. Patients with DLCO <80%.
* Group II Patients with DLCO≥80%.

Both groups will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years. The participant or his / her legal representative is willing and able to give informed consent to participate in the study.
* Female or male patients with age equal to or greater than 18 years.
* Smokers or ex-smokers with cumulative exposure ≥ 10 a / p
* Respiratory symptoms
* Normal spirometry.

Exclusion Criteria:

* Age under 18 years.
* Participation in another clinical study.
* Patients with a life expectancy of less than 2 years due to neoplasms or other serious systemic diseases.
* Refusal to sing informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 smokers or ex-smokers with cumulative exposure ≥ 10 a / p (years /pack) with respiratory symptoms presenting normal spirometry
Sampling Method: Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2021-09-10 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of Diffusion Capacity (DLCO) at 5 years | through study completion, an average of 5 years
  To determine the value of DLCO in COPD screening in smokers and ex-smokers with respiratory symptoms and normal spirometry (GOLD 0)

SECONDARY OUTCOMES:
Risk factors associated to the development of COPD | through study completion, an average of 5 years
  Risk factors associated to the development of COPD
Changes from baseline of inflammatory Markers at 2 and 5 years | 2 and 5 years
  To Study soluble receptors involved in inflammation processes and tissue repair in early disease stages.
Oxidative stress | through study completion, an average of 5 years
  To Study of oxidative stress parameters in early disease stages
Diffusion study | through study completion, an average of 5 years
  To Characterize patients in stage 0 of GOLD with impaired diffusion
Changes from baseline of High Resolution Computed Tomography (HRTC) at 5 years | Baseline and 5 years
  To determine changes in HRCT to identify subgroups of patients with different clinical and evolutionary trajectories
Airflow limitation Study | through study completion, an average of 5 years
  To Investigate the contribution of measuring lung volumes for the diagnosis of COPD when there is no evidence of airflow limitation in spirometry (GOLD 0).
Gender differences in value of diffusion (DLCO) | through study completion, an average of 5 years
  To assess if there are differences between men and women with diffusion disorder
Childhood background | Baseline
  To assess whether factors, such as the effect of lung development during childhood and adolescence, bronchial hyperreactivity and / or the role of infections influences the risk of developing the disease or its progression.
Comorbidity | through study completion, an average of 5 years
  To characterize the comorbidities associated with GOLD 0 patients and altered diffusion.

CONTACTS AND LOCATIONS:
Overall Officials: Cruz González, PhD, Study Director — Hospital Clínico Universitario de Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Valencia, Spain